CLINICAL TRIAL: NCT05824897
Title: The Cohort Study of the Correlation Between Serum 25(OH)D Level and Pregnancy Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aimin Zhao (Other)
Responsible Party: Sponsor-Investigator, Aimin Zhao, Chief physician, RenJi Hospital
Organization: RenJi Hospital (Other)
Other Study IDs: IIT-2023-0011
Record Dates: First submitted 2023-04-06; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Vitamin D Deficiency; Recurrent Miscarriage; Pregnancy Related
Keywords: vitamin D; pregnancy; recurrent spontaneous abortion
MeSH Terms: conditions — Vitamin D Deficiency; Abortion, Habitual; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Serum levels of vitamin D — Subjects in this study are grouped according to baseline serum levels of 25(OH)D. The serum level of total 25(OH)D ≥30ng/ml (75nM) is sufficient, 20-30ng/ml (50-75 nm) is insufficient, and less than 20ng/ml (50nM) is deficient.

SUMMARY:
The objective of this single-center prospective observational study is to clarify the trend of maternal serum 25(OH)D levels before pregnancy and during pregnancy, and to explore the correlation between serum 25(OH)D levels and subsequent pregnancy outcomes of patients with abortion, so as to provide certain scientific evidence for finding the optimal serum level of 25(OH)D and optimal vitamin D supplementation to maintain a healthy pregnancy.

DETAILED DESCRIPTION:
Women of reproductive age who meet the inclusion criteria are recruited from the outpatient department of Renji Hospital from November 2022 to December 2023. Subjects fill in the basic information at the outpatient clinic. After being included in the study, peripheral blood is collected before and during the first trimester (< 10 weeks), second trimester (22-24 weeks) and third trimester (32 weeks) to detect 25(OH)D, calcium, phosphorus and PTH levels. B-ultrasound examination is performed before pregnancy to record endometrial thickness, endometrial hemodynamic index (PI, RI and S/D) and uterine arterial hemodynamic index (PI, RI and S/D) during the luteal phase. Data are comprehensively analyzed through questionnaire form filling, laboratory examination, and clinical information records including pregnancy outcomes (final live birth rate, cesarean section rate, pregnancy loss rate, etc.), obstetric complications, and neonatal delivery information.

ELIGIBILITY:
Inclusion Criteria:

* ≥20 years old
* The chromosome karyotype of the couple is normal
* Color ultrasound examination results indicated that there was no organic disease related to reproductive tract
* No serious complications of surgery and medicine
* Agree and voluntarily sign informed consent

Exclusion Criteria:

* There are contraindications to pregnancy
* the initiative to give up pregnancy
* Severe medical and surgical complications, for example, liver disease was defined as serum alanine aminotransferase [ALT] or aspartic aminotransferase [AST]>3 x upper normal limit [ULN] after repeated testing
* Concomitant malignant tumor, malignant tumor developed in the last 5 years (except for the skin squamous basal cell carcinoma that has been removed and considered cured). Subjects who developed malignant tumors more than 5 years ago should provide evidence of remission or cure. Subjects with a history of cervical cancer were eligible if they could demonstrate that their cervical cancer had been cone removed or cured within the past 3 years
* Known human immunodeficiency virus (HIV) positive and/or hepatitis B surface antigen or hepatitis C virus antibody positive at screening visit
* With a history of chronic infections such as mycoplasma, chlamydia, cryptococcus, and invasive fungal infections should be discussed with the principal investigator

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women of childbearing age
Study Population: Women of childbearing age who are ready to become pregnant or already pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
pregnancy loss | Up to 28 weeks
  After a positive urinary hCG pregnancy test at home or clinically, there were no clinical signs of pregnancy on subsequent ultrasound or signs of pregnancy were lost after ultrasound confirmation.

SECONDARY OUTCOMES:
Live birth | Up to 20 weeks
  A live baby born after 23 weeks of gestation
Premature birth | 9 weeks
  Delivery between 28 and 37 weeks gestation
Preeclampsia | 20 weeks
  New hypertension (blood pressure greater than 140/90 mmHg) after 20 weeks of gestation combined with new unexplained urinary protein greater than or equal to 300mg/24h or a urinary protein/creatinine ratio greater than or equal to 0.3 or other conditions
Gestational diabetes mellitus | 4 weeks
  Perform a 75-g OGTT with plasma glucose measurement when patient is fasting and at 1 and 2 h, at 24-to-28-wk gestation in women not previously diagnosed with overt diabetes
  The diagnosis of GDM is made when any one of the following plasma glucose values are met or exceeded:
  Fasting: 92 mg/dL
  1. h: 180 mg/dL
  2. h: 153 mg/dL
Fetal growth restriction | Up to 28 weeks
  Fetal weight below the 10th percentile of the mean weight for its gestational age or below 2 standard deviations of the mean weight

CONTACTS AND LOCATIONS:
Overall Officials: Aimin Zhao, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No